CLINICAL TRIAL: NCT03276611
Title: Assessment of Pulmonary Artery Pressure and Right Sided Hemodynamics in Patients With OSA Before and After CPAP TTT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yahia Shabeeb Fadel Madi, principle investigator, Assiut University
Other Study IDs: 17100139
Record Dates: First submitted 2017-08-21; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: Assessment; pulmonary; artery; right; sided; hemodynamics; patients; sleep; apnea; syndrome; contionous; positive; air; way; pressure; treatment
MeSH Terms: conditions — Apnea; Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: echocardiograghy — transthoracic echocardiograghy

SUMMARY:
Obstructive sleep apnea (OSA) is a frequent sleep-related breathing disorder with an incidence of 5-20% in the middle-aged population in Europe and Northern America . plumonary hypertension is present in 12%-34% of patients with osa.continous positive air way pressureis the main standard treatment ofOSA.Echocardiograghy is the most common non invasive imaging method for assessment the effect on right ventricular function.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a frequent sleep-related breathing disorder with an incidence of 5-20% in the middle-aged population in Europe and Northern America . Pathophysiologic consequences of OSA are increased sympathetic activity, hypoxia, hypercapnia, increased left ventricular after-load , acute arterial hypertension, increased diastolic and systolic pressure of the right ventricle, atrial dilation. Recent studies have shown that OSA is an independent risk factor for cardiovascular mortality and morbidity. OSA has a social impact because of fragmentation of sleep leads to increased daytime sleepiness, decreased intellect, behavioral and personality changes, enuresis and sexual dysfunction.

Pulmonary hypertension is present in 12%-34% of patients with Obstructive Sleep Apnea syndrome. When PH occurs as a consequence of OSA however symptoms may not be present because of obesity and alack of physical exertion or symptoms of PH may be overlapped by other cardiovascular abnormalities.

Continuous positive air way pressure therapy is the main standard treatment of OSA works the best in the most people as positive pressure ventilation functions as a pneumatic splint for the collapsing upper air way. Echocardiography is the most common non invasive imaging method for assessment the effect of right ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* Moderate and severe OSA and candidates for initiation of CPAP therapy.

Exclusion Criteria:

* Significant lung disease ,lfet sided heart failure,end stage malignancy and advanced organ failure.

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients will be evaluated at the sleep lap of chest department of assiut university hospital over 1 year will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of OSA and CPAP therapy on pulmonary artery pressure and right sided hemodynamics | Transthoracic echocardiography will be planned for evaluation of OSA patients regularly used CPAP (at least 5hrs/night) before and after 3 month of initiation of CPAP therapy.
  Transthoracic echocardiography to determine right ventricle and right atrium functional parameters and dimensions and pulmonary artery systolic pressure, echocardiography will be planned for evaluation of OSA before initiation of CPAP therapy and after 3 month of CPAP therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yahia Shabeeb, MBBCH, Principal Investigator — Assiut University
Locations (1):
- Amr Youssef, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park JG, Ramar K, Olson EJ. Updates on definition, consequences, and management of obstructive sleep apnea. Mayo Clin Proc. 2011 Jun;86(6):549-54; quiz 554-5. doi: 10.4065/mcp.2010.0810. PMID 21628617
- [Background] Gottdiener JS, Bednarz J, Devereux R, Gardin J, Klein A, Manning WJ, Morehead A, Kitzman D, Oh J, Quinones M, Schiller NB, Stein JH, Weissman NJ; American Society of Echocardiography. American Society of Echocardiography recommendations for use of echocardiography in clinical trials. J Am Soc Echocardiogr. 2004 Oct;17(10):1086-119. doi: 10.1016/j.echo.2004.07.013. No abstract available. PMID 15452478
- [Background] Kim SH, Cho GY, Shin C, Lim HE, Kim YH, Song WH, Shim WJ, Ahn JC. Impact of obstructive sleep apnea on left ventricular diastolic function. Am J Cardiol. 2008 Jun 1;101(11):1663-8. doi: 10.1016/j.amjcard.2008.01.056. Epub 2008 Apr 18. PMID 18489948
- [Background] Jurcut R, Giusca S, La Gerche A, Vasile S, Ginghina C, Voigt JU. The echocardiographic assessment of the right ventricle: what to do in 2010? Eur J Echocardiogr. 2010 Mar;11(2):81-96. doi: 10.1093/ejechocard/jep234. Epub 2010 Feb 2. PMID 20124362
- Available data/document: Statistical Analysis Plan — http://www.ncbi.nlm.nih.gov/